CLINICAL TRIAL: NCT06650683
Title: Impact of Providing Nursing Support on Parental Stress Related to Preoperative Care of a Newborn with Hirschsprung's Disease
Acronym: HirscHAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCAPHM22_0037; 2022-A02696-37 (Other: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Hospitalisation at Home (HAH) (Experimental): families living in Marseille, whose parents will be able to return home under the supervision of nursery nurses from the pediatric HAH.
  Interventions: Behavioral: Pediatric HAH
- Without Hospitalisation at Home (HAH) (No Intervention): Families living outside Marseille whose parents will have to carry out nursings at home independently, without the help of pediatric HAH.

INTERVENTIONS:
Behavioral: Pediatric HAH — Pediatric HAH nursing support for home nursery care provided by parents as part of their child's disease.
  Arms: With Hospitalisation at Home (HAH)

SUMMARY:
Impact of providing nursing support on parental stress related to preoperative care of a newborn with Hirschsprung's disease

ELIGIBILITY:
Inclusion Criteria:

* Families (one or two parents) with a newborn or infant under 2 months with confirmed or suspected Hirschsprung disease, for whom nursings are effective and performed 1 to 2 times a day while waiting for surgery.
* With a possible return home before surgery
* With an information leaflet and non-opposition form signed by one or both parent(s) or by the legal representative.

Exclusion Criteria:

* The absence of daily nursings
* Initial ineffectiveness of nursings requiring a digestive stoma
* Failure to return home before surgery
* Refusal of one or both parent(s) or legal representative(s)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Questionnary to evaluate stress on parents | From enrollment to the end of treatment at 6 months
  Evaluation of the impact on parental stress of nursing support by pediatric HAH in nursery care performed at home by parents as part of their child with Hirschsprung using Perinatal Posttraumatic Stress Disorder Questionnaire (PPQ).

SECONDARY OUTCOMES:
Auto-Questionnary MIB (Mother Infant Bounding) to evaluate the impact of nursing support | From enrollment to the end of treatment at 6 months
  Estimate the impact of nursing support by pediatric HAH in nursery care performed at home by parents on the development of the parent-child bond, the burden felt by parents in relation to their child's illness, the length of pre-operative hospital stay (initial and re-hospitalization), the pre-operative complications (recurrent occlusion, enterocolitis) and the home nursing care provided by parents (quality of nursings, pace of nursings, difficulties encountered, child's tolerance)
Self-Questionnary Burden inventory to evaluate the nursery training provided | From enrollment to the end of treatment at 6 months
  Evaluate nursery training provided by the paramedical team (feedback from parents) : parent training (nursing, understanding illness, understanding illness-related risks) and training aids (sheet, video)

CONTACTS AND LOCATIONS:
Locations (1):
- APHM, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided